## 高醫/大同骨科 rotator cuff lesions 病人日誌

## Visit 1

| Genera | al and preoperative data: |
|--------|-------------------------------------------------------------|
| 0 | Chart number: |
| 0 | Name: |
| 0 | ICF signed date: |
| 0 | MRI examination date: |
| 0 | Echo examination date: |
| 0 | Age: |
| 0 | Gender:malefemale |
| 0 | Phone number: |
| 0 | BMI: |
| 0 | Occupation: |
| 0 | Smoking:noyes,ppd foryears |
| 0 | Dominant hand: |
| 0 | Affected hand: |
| 0 | Symptom duration:months |
| 0 | underlying disease: nil |
| | ☐ Diabetes ☐ RA ☐ breast CA s/p OP ☐ Thyroid disease |
| | others: |
| 0 | Previous conservative treatment: |
| | ☐Warm packing/Wax therapy ☐Immobilization ☐TENS ☐ultrasound |
| | Local injection Acupuncture others: |
| 0 | medication list: |
| Record | date: Recorder: |

版本:1 版本日期: 2023 年 08 月 23 日

| Visit 2 | |
|-----------------|----------------------------------------------------|
| Treatment data: | |
| 0 | Treatment date: |
| 0 | Random group: |
| 0 | VAS: |
| 0 | Constant-Murley Shoulder Score (CMSS) : |
| 0 | American Shoulder and Elbow Surgeons (ASES) Score: |
| 0 | Shoulder joint activities: |
| 0 | Blood:ml |
| 0 | Anesthesia: |
| 0 | Treatment hand: |
| 0 | Treatment duration(注射時間): min |

Recorder:

Record date:

版本:1 版本日期: 2023 年 08 月 23 日

Visit 3
Postop

| Postop | perative 4-week follow-up: |
|---------|----------------------------------------------------|
| 0 | VAS: |
| 0 | Constant-Murley Shoulder Score (CMSS) : |
| 0 | American Shoulder and Elbow Surgeons (ASES) Score: |
| 0 | Shoulder joint activities: |
| 0 | Complication: (可複選) |
| | Superficial infection |
| | Deep infection |
| | • Allergy |
| | • |
| | • scar hypertrophy |
| | Scar hypersensitivity |
| | <ul> <li>secondary operation</li> </ul> |
| | •other: |
| 0 | 備註(AE): |
| Record | date: |
| Visit 4 | |
| Postop | perative 12-week follow-up: |
| 0 | VAS: |
| 0 | Constant-Murley Shoulder Score (CMSS) : |
| 0 | American Shoulder and Elbow Surgeons (ASES) Score: |
| 0 | Shoulder joint activities: |
| 0 | Complication: (可複選) |
| | Superficial infection |
| | Deep infection |
| | <ul> <li>Allergy</li> </ul> |
| | <ul><li>■ pillar pain</li></ul> |
| | • scar hypertrophy |
| | Scar hypersensitivity |
| | secondary operation |
| | •other: |
| 0 | 備註(AE): |
| Record | l date: Recorder: |

版本:1 版本日期: 2023 年08 月23 日

## Visit 5

## Postoperative 24-week follow-up:

| VAS: |
|----------------------------------------------------|
| Constant-Murley Shoulder Score (CMSS) : |
| American Shoulder and Elbow Surgeons (ASES) Score: |
| Shoulder joint activities: |
| Complication: (可複選) |
| Superficial infection |
| Deep infection |
| • Allergy |
| • |
| • scar hypertrophy |
| Scar hypersensitivity |
| secondary operation |
| •other: |
| Echo: |
| 備註(AE): |
| date: |

版本:1 版本日期: 2023 年 08 月 23 日